CLINICAL TRIAL: NCT04471558
Title: Evaluation of the Effect of Music on Young Practitioner's Stress During Endodontic Treatment
Brief Title: Effect of Music on Young Practitioner's Stress During Endodontic Treatment
Acronym: MUSIQUENDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: MUSIQUENDO (29BRC20.0045)
Record Dates: First submitted 2020-07-02; First posted 2020-07-15 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Endodontic Disease
Keywords: Root canal treatment; Music
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Music Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Music group: A part of the care is realized with music.
  Interventions: Other: Music
- Control group: The entire care is realized without music.

INTERVENTIONS:
Other: Music — A part of the RCT will be performed with music in the room. The music will be switch on just before anesthesia and off after the postoperative rest.
  Groups: Music group

SUMMARY:
According to several studies, patients consider endodontic treatment as one of the most stress-inducing dental procedures. Two studies demonstrated that music enables the patient to be less stressed during RCT.

RCTs are also stressful for the practitioner, and particularly for students who start their dental practice. Endodontic and prosthetic cares are considered the most demanding by students. RCT requires high degree of precision in gestures and patience because those technical acts are, in part, blindly realised and can be long. In a preliminary study, it was found that the most stress-inducing steps for the students during endodontic treatment are root-canal preparation and filling.

The beneficial side of listening to music on the patient's stress during RCT has been proved; but to our knowledge, no study assessed the effect of listening to music on the stress of the practitioner and more particularly of the young practitioner, during endodontic treatment, and in particular during root canal preparation. This is the main aim of this study.

DETAILED DESCRIPTION:
Root canal treatment (RCT) consists in eliminating infected and /or inflammatory tissues inside the root canal system of the tooth by a chemo-mechanical preparation and then filling the latter in a three-dimensional, bacteriostatic and durable way to enable healing. This treatment is commonly carried out and can sometimes be long and tedious, as, for instance, on molars with several roots.

According to numerous studies, patients consider endodontic treatment as one of the most stress-inducing dental procedures. The preliminary study Stressendo has shown that anesthesia is the most stressful step for the patient. In some studies, patients also fear the pain and discomfort during RCT. Stress and pain have neurological consequences including the activation of neuroendocrine system which secretes catecholamines. Those act on the heart by increasing the heart rate and arterial pressure.

Two studies demonstrated that relaxing music enables the patient to be less stressed during RCT.

Another study has shown that music also enables the patient to feel less painful during dental care. This would be explained by the fact that music can help reducing the sound perceived as stressful for the patients, in addition to the distraction it produces. Music also has a physiological and psychological role, which enables the patient to feel more relaxed. However, it would depend on its style and the fact that the patient likes it or not. Many studies demonstrated that when the patient likes the music used, the reduction of anxiety is higher than with relaxing music.

RCTs are stressful for the patient, but one must keep in mind that it is also stressful for the practitioner, and particularly for students who start their dental practice.

The students have to treat patients with many parameters to manage. Combining theoretical and clinical practice knowledge is difficult and stressful for students according to a study. Endodontic and prosthetic cares are considered the most demanding by students. RCT requires high degree of precision in gestures and patience because those technical acts are, in part, blindly realised and can be long. In a preliminary study, it was found that the most stress-inducing steps for the students during endodontic treatment are root-canal preparation and obturation.

The beneficial side of listening to music (relaxing music) on the patient's stress during RCT has been proved; but to our knowledge, no study assessed the effect of listening to appreciated music on the stress of the practitioner and more particularly of the young practitioner, during endodontic treatment and in particular root canal preparation.This is the main aim of this study.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* person between 18 and 70 years old
* patient who needs an endodontic treatment on a molar tooth
* person affiliated to or beneficiary of a social security scheme
* patient consent

Student:

* 4th, 5th or 6th year student in odontology
* student consent
* student affiliated or beneficiary of a social security scheme

Exclusion Criteria:

Patients and students:

* Pregnant woman
* Major protected by law
* Non-cooperating person who does not speak or read French fluently, or unable to understand the principle of a stress scale and unable to collaborate on tests.
* Person with a psychiatric diagnosis of schizophrenia, delusional disorders and other personality disorders (ICD-10: F20 to F29; DSM IV: Axis II)
* Person with a pathology that does not allow interpretation of cardiovascular results (heart rhythm disorders, hypertension)
* A person taking medication that affects the heart rate (antiarrhythmics, antihypertensives, beta blockers, etc.).
* Refusal to participate
* Hearing impaired person who does not perceive sounds correctly
* Hearing aid wearer
* Person who has already participated in this protocol

Patient:

* Patient at high risk of infective endocarditis (necrotic pulp)
* Patient whose tooth has no functional future and cannot be permanently restored
* Patient whose tooth has insufficient periodontal support

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient who needs an endodontic treatment and his practionner.
Sampling Method: Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-12-09 (Estimated); Study Completion 2022-12-09 (Estimated)

PRIMARY OUTCOMES:
Change in practitioner's stress during canal root preparation | T1bis (preoperative step of the second session of RCT); T4 (canal root preparation)
  The student will evaluate his stress on an Analogic Visual Scale (AVS). 0 is "very relax" and 10 is "extremely stressed"

SECONDARY OUTCOMES:
Variation of the practitioner's stress at different stages. | Each step of the RCT
  The student will evaluate his stress on an Analogic Visual Scale (AVS). 0 is "very relax" and 10 is "extremely stressed". AVS will be compared between each step and the preoperative step of the corresponding session. We will also compare the 3 preoperative steps and the 2 anesthesia steps.
Variation of the patient's stress at different stages. | Each step of the RCT
  The patient will evaluate his stress on an Analogic Visual Scale (AVS). 0 is "very relax" and 10 is "extremely stressed". AVS will be compared between each step and the preoperative step of the corresponding session. We will also compare the 3 preoperative steps and the 2 anesthesia steps.
Variation of the patient's pain at different stages. | Each step of the RCT
  The patient will evaluate his pain on an Analogic Visual Scale (AVS). 0 is "no pain" and 10 is "extremely painful". AVS will be compared between each step and the preoperative step of the corresponding session. We will also compare the 3 preoperative steps and the 2 anesthesia steps.
Variation of the patient's discomfort at different stages. | Each step of the RCT
  The patient will evaluate his discomfort on an Analogic Visual Scale (AVS). 0 is "very comfortable" and 10 is "extremely uncomfortable". AVS will be compared between each step and the preoperative step of the corresponding session. We will also compare the 3 preoperative steps and the 2 anesthesia steps.
Relation between patient and student's stress | Each step of the RCT
  The patient and student will evaluate their stress on an Analogic Visual Scale (AVS). 0 is "very relax" and 10 is "extremely stressed".
Evaluate the stress induced by an RCT with Spielberger's questionaires | Day 0, Day 15, Day 30
  Spielberger's questionnaires Y1 and Y2 for anxiety evaluation will be done on both patients and students to evaluate their general (Y2) and induced (Y1) anxiety. Both questionnaires are composed of 20 questions, total score is between 0 and 80. The higher the score, the more anxious the person is.
Dental anxiety | Day 0
  Dental anxiety will be evaluated by the Dental Anxiety Scale of Corah which consist of 4 questions. The total score is calculated between 4 and 20. The highest the score, the more anxious the person is.
Patient's blood pressure | Each step of the RCT
  Patient's systolic and diastolic blood pressure will be evaluated at each stage of the RCT, with a tensiometer (mmHg). This parameter can reflect the stress.
Patient's heart rate | Each step of the RCT
  Patient's heart rate will be evaluated at each stage of the RCT, with a cardiofrequencemeter (number of pulses per minute). This parameter can reflect the patient's stress.
Patient's heart rate variability | during the RCT (day 0 and day 15)
  Patient's heart rate variability will be evaluated during the RCT, with a cardiofrequencemeter (ms). This parameter can reflect the patient's stress.
Student's blood pressure | Each step of the RCT
  Student's systolic and diastolic blood pressure will be evaluated at each stage of the RCT, with a tensiometer (mmHg). This parameter can reflect the stress.
Student's heart rate | Each step of the RCT
  Student's heart rate will be evaluated at each stage of the RCT, with a cardiofrequencemeter (number of pulses per minute). This parameter can reflect the student's stress.
Student's heart rate variability | during the RCT (day 0 and day 15)
  Student's heart rate variability will be evaluated during the RCT, with a cardiofrequencemeter (ms). This parameter can reflect the student's stress.
Musical training questionnaire | Day 0
  An identical questionnaire for the practitioner and the patient will be filled for the music group. It aims to assess their musical training/knowledge and to evaluate whether a musical training/knowledge has an impact on the effect of the music during the RCT.
patient's satisfaction assessed by a scale and a questionnaire | Day 15
  The patient will assess his satisfaction on an Analogic Visual Scale (AVS). 0 is "not satisfied" and 10 is "extremely satisfied". The questionnaire aims at determining the sources of satisfaction.
student's satisfaction assessed by a scale and a questionnaire | Day 15
  The student will assess his satisfaction on an Analogic Visual Scale (AVS). 0 is "not satisfied" and 10 is "extremely satisfied". The questionnaire aims at determining the sources of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending five years following the final study report completion.
Access Criteria: Data access request will be reviewed by the internal committee of Brest University Hospital. Requestor will be required to sign and complete a data access agreement.